CLINICAL TRIAL: NCT07049302
Title: Comparison of Conventional and Non-Conventional Cardiovascular Risk Factors and Their Association With Acute Coronary Syndrome
Brief Title: Comparison of Conventional and Non-Conventional CRF and Their Association With Acute Coronary Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/911
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Coronary Syndrome
MeSH Terms: conditions — Angina, Unstable

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional Risk Factor Assessment
  Interventions: Combination Product: Conventional Risk Factor Assessment
- Non-Conventional Risk Factor
  Interventions: Combination Product: Non-Conventional Risk Factor

INTERVENTIONS:
Combination Product: Conventional Risk Factor Assessment — Participants in Group 1 will undergo evaluation for conventional cardiovascular risk factors associated with Acute Coronary Syndrome (ACS
  Groups: Conventional Risk Factor Assessment
Combination Product: Non-Conventional Risk Factor — Participants in Group 2 will be assessed for non-conventional cardiovascular risk factors associated with Acute Coronary Syndrome (ACS).
  Groups: Non-Conventional Risk Factor

SUMMARY:
This research aims to compare conventional and non-conventional cardiovascular risk factors and their association with Acute Coronary Syndrome (ACS). Conventional risk factors such as hypertension, diabetes mellitus, dyslipidemia, smoking, and family history are well-established contributors to ACS. However, emerging non-conventional risk factors-including elevated inflammatory markers , homocysteine levels, lipoprotein(a), psychological stress, and lifestyle factors-are gaining attention for their potential role in cardiovascular events.

DETAILED DESCRIPTION:
The study will involve a cross-sectional analysis of ACS patients, examining the prevalence and impact of both types of risk factors. By assessing their relative contributions, the study aims to enhance understanding of ACS pathogenesis, identify at-risk populations more accurately, and support more comprehensive prevention strategies. The findings may help broaden clinical risk assessment tools and guide personalized interventions to reduce the incidence of ACS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with ACS.
* Patients providing informed consent for participation.

Exclusion Criteria:

* Patients with chronic heart diseases unrelated to ACS.
* Patients unable to provide consent due to critical illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will involve a cross-sectional analysis of ACS patients, examining the prevalence and impact of both types of risk factors. By assessing their relative contributions, the study aims to enhance understanding of ACS pathogenesis, identify at-risk populations more accurately, and support more comprehensive prevention strategies. The findings may help broaden clinical risk assessment tools and guide personalized interventions to reduce the incidence of ACS.
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Structured Smoking Questionnaire | 12 Months
  A structured smoking questionnaire is a tool used to assess an individual's smoking habits, level of nicotine dependence, and potential motivations for smoking. These questionnaires typically include questions about cigarette consumption, brand preferences, smoking patterns, and the perceived effects of smoking.
  nterpretation: Higher scores indicate greater nicotine dependence.
  Scores:
  0-2: Very low dependence 3-4: Low dependence 5: Moderate dependence 6-7: High dependence 8-10: Very high dependence

CONTACTS AND LOCATIONS:
Locations (1):
- Tertiary care hospital, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No